CLINICAL TRIAL: NCT01287741
Title: A Phase III, Multicenter, Open-Label Randomized Trial Comparing the Efficacy of GA101 (RO5072759) in Combination With CHOP (G-CHOP) Versus Rituximab and CHOP (R-CHOP) in Previously Untreated Patients With CD20-Positive Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: A Study of Obinutuzumab in Combination With CHOP Chemotherapy Versus Rituximab With CHOP in Participants With CD20-Positive Diffuse Large B-Cell Lymphoma (GOYA)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was closed by the Sponsor according to the protocol-specified minimum post-treatment follow-up period of 3 years.
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO21005; 2010-024194-39
Record Dates: First submitted 2011-01-31; First posted 2011-02-01 (Estimated); Results first posted 2017-08-17 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; obinutuzumab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

ARMS (2):
- Rituximab+Chemotherapy (Active Comparator): Participants received eight 21-day cycles of rituximab, combined with six or eight cycles of standard cyclophosphamide, doxorubicin, vincristine, and prednisone/prednisolone (CHOP) chemotherapy (21-day cycles). Prior to study start, study centers chose whether they planned to administer 6 or 8 cycles of CHOP chemotherapy.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone
- Obinutuzumab+Chemotherapy (Experimental): Participants received eight 21-day cycles of obinutuzumab, combined with six or eight cycles of standard cyclophosphamide, doxorubicin, vincristine, and prednisone/prednisolone (CHOP) chemotherapy (21-day cycles). Participants received an additional two doses of obinutuzumab on Days 8 and 15 of Cycle 1. Prior to study start, study centers chose whether they planned to administer 6 or 8 cycles of CHOP chemotherapy.
  Interventions: Drug: Obinutuzumab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Rituximab — Rituximab at a dose of 375 mg/m^2, administered by intravenous (IV) infusion on Day 1 of each 21-day cycle for 8 cycles.
  Other Names: MabThera, Rituxan
  Arms: Rituximab+Chemotherapy
Drug: Obinutuzumab — Obinutuzumab 1000 mg IV infusion, administered on Day 1 of each 21-day cycle for 8 cycles. During Cycle 1, obinutuzumab was also infused on Days 8 and 15.
  Other Names: GA101, RO5072759
  Arms: Obinutuzumab+Chemotherapy
Drug: Cyclophosphamide — Cyclophosphamide 750 milligrams per square metre (mg/m^2), administered intravenously (IV) on Day 1 of each 21-day cycle.
Drug: Doxorubicin — Doxorubicin 50 mg/m^2 IV, administered on Day 1 of each 21-day cycle.
Drug: Vincristine — Vincristine 1.4 mg/m^2 (maximum 2 mg) IV, administered on Day 1 of each 21-day cycle.
Drug: Prednisone — Prednisone 100 mg (or equivalent prednisolone or methylprednisolone), administered orally on Days 1-5 of each 21-day cycle.

SUMMARY:
This open-label, randomized, parallel group study will evaluate the efficacy and safety of obinutuzumab in combination with cyclophosphamide, doxorubicin, vincristine, and prednisolone or prednisone (CHOP) chemotherapy versus rituximab (MabThera/Rituxan) with CHOP in previously untreated participants with cluster of differentiation 20 (CD20)-positive diffuse large B-cell lymphoma (DLBCL). Participants will be randomized to receive either obinutuzumab 1000 milligrams (mg) intravenously (IV) every 21 days or rituximab 375 milligrams per square meter (mg/m^2) IV every 21 days for 8 cycles, in addition to 6-8 cycles of CHOP chemotherapy IV every 21 days. Participants randomized to the obinutuzumab arm will receive an additional two doses on Days 8 and 15 of Cycle 1. Anticipated time on study treatment is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated CD20-positive DLBCL
* At least 1 bi-dimensionally measurable lesion (greater than [>]1.5 centimeters [cm] in its largest dimension on the computed tomography [CT] scan)
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Adequate hematological function
* Low-intermediate, high-intermediate or high-risk International Prognostic Index (IPI) score (low-risk IPI score: IPI 1 irrespective of bulky disease or IPI 0 with bulky disease, defined as one lesion greater than equal to (>/=) 7.5 cm)
* Left ventricular ejection fraction (LVEF) >/=50 percent (%) on cardiac multiple-gated acquisition (MUGA) scan or cardiac echocardiogram

Exclusion Criteria:

* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products or to any component of CHOP or obinutuzumab
* Contraindication to any of the individual components of CHOP, including prior receipt of anthracyclines
* Participants with transformed lymphoma and participants with follicular lymphoma IIIB
* Prior therapy for DLBCL, with the exception of nodal biopsy or local irradiation
* Prior treatment with cytotoxic drugs or rituximab for another condition (for example, rheumatoid arthritis) or prior use of an anti-CD20 antibody
* Prior use of any monoclonal antibody within 3 months of the start of Cycle 1
* Corticosteroid use of >30 milligrams per day (mg/day) of prednisone or equivalent, for purposes other than lymphoma symptom control
* Primary central nervous system (CNS) lymphoma and secondary CNS involvement by lymphoma, mantle-cell lymphoma (MCL), or histologic evidence of transformation to a Burkitt lymphoma, primary mediastinal DLBCL, primary effusion lymphoma, plasmablastic lymphoma, and primary cutaneous DLBCL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1418 (Actual)
Dates: Start 2011-07-26 (Actual); Primary Completion 2016-04-29 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (235):
- United States (36):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Ironwood Cancer TX & Rsch Ctrs, Chandler, Arizona
  - Arizona Oncology, Tucson, Arizona
  - California Cancer Associates for Research & Excellence, Inc., Encinitas, California
  - cCare, Encinitas, California
  - UCLA - School of Medicine; Division of Hematology/Oncology, Los Angeles, California
  - Rocky Mountain Cancer Center - Aurora, Aurora, Colorado
  - Florida Cancer Specialists; Department of Oncology, Fort Myers, Florida
  - Florida Cancer Specialists; Saint Petersburg, St. Petersburg, Florida
  - Central Georgia Cancer Care PC, Macon, Georgia
  - Illinois Cancer Care, P.C. - Galesburg, Galesburg, Illinois
  - Joliet Oncology-Hematology; Associates, Ltd., Joliet, Illinois
  - Cancer Care & Hematology; Specialists of Chicagoland, Niles, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Mercy Oncology / Hematology Center; Oncology, Portland, Maine
  - Park Nicollet Clin-Cancer Ctr, Saint Louis Park, Minnesota
  - Minnesota Oncology Hematology Woodbury, Woodbury, Minnesota
  - New York Oncology Hematology, P.C., Albany, New York
  - Mecklenburg Medical Group Charlotte, Charlotte, North Carolina
  - Forsyth Regional Cancer Center; Piedmont Hematology/Oncology Associates, Winston-Salem, North Carolina
  - Signal Point Clinical; Research Center, LLC, Middletown, Ohio
  - Cleveland CL N Coast Cancer Cr, Sandusky, Ohio
  - Willamette Valley Cancer Insitute and Research Center, Springfield, Oregon
  - Medical University of SC (MUSC), Charleston, South Carolina
  - South Carolina Oncology Associates - SCRI, Columbia, South Carolina
  - Chattanooga Oncology and Hematology Associates, PC, Chattanooga, Tennessee
  - Tennessee Onc., PLLC - SCRI, Nashville, Tennessee
  - Texas Oncology, Pa - Amarillo, Amarillo, Texas
  - Texas Oncology-Fort Worth 12th Ave, Fort Worth, Texas
  - MD Anderson Cancer Center Department of Lymphoma & Myeloma, Houston, Texas
  - Cancer Care Centers of South Texas-HOAST - San Antonio, New Braunfels, Texas
  - Virginia Cancer Institute, Richmond, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - Virginia Cancer Specialists - Winchester, Winchester, Virginia
  - Northwest Medical Specialties, Tacoma, Washington
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington
- Argentina (3):
  - Instituto Damic, Córdoba
  - Sanatorio Britanico: Hematologia, Rosario
  - Sanatorio Parque de Rosario, Rosario
- Australia (4):
  - Cairns Base Hospital; Cancer Care Centre, Cairns, Queensland
  - Frankston Hospital; Oncology/Haematology, Frankston, Victoria
  - Monash Medical Centre; Haematology, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (3):
  - Tiroler Landeskrankenanstalten Ges.M.B.H.; Innere Medizin Abt. Für Hämatologie & Onkologie, Innsbruck
  - Lkh Salzburg - Univ. Klinikum Salzburg; Iii. Medizinische Abt., Salzburg
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin I - Hämatologie & Hämostaseologie, Vienna
- Brazil (5):
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas Oncologicas - CEPON, Florianópolis, Santa Catarina
  - Instituto de Ensino e Pesquisa Sao Lucas - IEP, São Paulo, São Paulo
  - Hospital Santa Marcelina;Oncologia, São Paulo, São Paulo
- Canada (15):
  - Tom Baker Cancer Centre; Dept of Medicine, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre; Oncology, Halifax, Nova Scotia
  - Ottawa General Hospital, Ottawa, Ontario
  - North York General Hospital, Toronto, Ontario
  - Humber River Hospital, Toronto, Ontario
  - University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario
  - Hopital Maisonneuve- Rosemont; Oncology, Montreal, Quebec
  - Chum Hopital Notre Dame; Centre D'Oncologie, Montreal, Quebec
  - Mcgill University - Royal Victoria Hospital; Oncology, Montreal, Quebec
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec
  - Hopital de L'Enfant-Jesus; Hematology, Québec, Quebec
  - Centre de sante et de services sociaux Rimouski Neigette, Rimouski, Quebec
  - Saskatoon Cancer Centre; Uni of Saskatoon Campus, Saskatoon, Saskatchewan
- China (28):
  - Cancer Hospital Chinese Academy of Medical Sciences., Beijing
  - Peking University First Hospital, Beijing
  - The Affiliated Hospital of Military Medical Sciences(The 307th Hospital of Chinese PLA), Beijing
  - Beijing Cancer Hospital, Beijing
  - Beijing Hospital of Ministry of Health; Hematology, Beijing
  - General Hospital of Chinese PLA; Department of Hematology, Beijing
  - the First Hospital of Jilin University, Changchun
  - Hu Nan Provincial Cancer Hospital, Changsha
  - Fujian Medical University Union Hospital, Fujian
  - Fujian Cancer Hospital, Fuzhou
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Guangdong General Hospital, Guangzhou
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The Second Affiliated Hospital to Nanchang University, Nanchang
  - Jiangsu Cancer Hospital, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - The First Affiliate Hospital of Guangxi Medical University, Nanning
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Changhai Hospital of Shanghai, Shanghai
  - First Hospital of China Medical University, Shenyang
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Cancer Hospital, Tianjin
  - Xiehe Hospital, Tongji Medical College Huazhong University of Science & Technology, Wuhan
  - Union Hospital of Tongji Medical College, Dept. of Cancer Center; Cancer Center, Wuhan
  - The Second Affiliated Hospital of The Fourth Military Medical University (Tangdu Hospital), Xi'an
- Colombia (3):
  - Fundacion Cardioinfantil, Bogotá
  - Organizacion Sanitas Internacional, Bogotá
  - FOSCAL, Floridablanca
- Czechia (3):
  - Fakultni nemocnice Brno; Interni hematologicka a onkologicka klinika, Brno
  - Fn Hr. Kralove; IV. Interni Hematologicka Klinika, Hradec Králové
  - Vseobecna Fakultni Nemocnice v Praze, I. Interni Klinika - Klinika Hematoonkologie VFN a 1. LF UK, Prague
- Denmark (3):
  - Aarhus Universitetshospital, Hæmatologisk Afdeling R, Aarhus
  - Rigshospitalet; Hæmatologisk Klinik, København Ø
  - Sygehus Syd Roskilde; Onkologisk/haematologisk ambulatorium, Roskilde
- Germany (7):
  - Uniklinik RWTH Aachen; Klinik IV; Klinik Hämatologie, Onkologie, Hämostaseologie und Stammz, Aachen
  - Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin
  - Universitätsklinikum "Carl Gustav Carus"; Medizinische Klinik und Poliklinik I, Dresden
  - Friedrich-Alexander-Universität Erlangen-Nürnberg; Medizinische Klinik V, Erlangen
  - Klinik der Justus-Liebig-Universität; Innere Medizin, Giessen
  - Uniklinik Heidelberg, Medizinische Klinik & Poliklinik V, Heidelberg
  - Universitätsklinikum Würzburg; Medizinische Klinik und Poliklinik II; Hämatologie / Onkologie, Würzburg
- Hong Kong (2):
  - Pamela Youde Nethersole Eastern Hospital; Department of Medicine, Hong Kong
  - Queen Mary Hospital; Dept of Medicine, Hong Kong
- Hungary (7):
  - Semmelweis University, First Dept of Medicine, Budapest
  - National Institute of Oncology, A Dept of Internal Medicine, Budapest
  - University of Debrecen Medical and Health Science Center, Institute of Internal medicine Building B, Debrecen
  - Petz Aladar Megyei Korhaz; Hematologia, Győr
  - Kaposi Mor Teaching Hospital, Dept of Internal Medicine/Hematology, Kaposvár
  - University of Pecs, I st Dept of Internal Medicine, Pécs
  - University of Szeged, II Dept of Internal Medicine, Szeged
- Italy (31):
  - Uni Degli Studi Di Bari, Policlinico; Cattedra Di Ematologia,Dipart. Di Medicina Interna E Publica, Bari, Apulia
  - IRCCS Ospedale Casa Sollievo Della Sofferenza; Ematologia E Trapianto Di Midollo Osseo, San Giovanni Rotondo, Apulia
  - Az. Osp. C. Panico; Rep. Ematologia E Trapianto, Tricase - LE, Apulia
  - Ospedale Riuniti; Divisione Di Ematologia, Reggio Calabria, Calabria
  - Istituto Nazionale Tumori Irccs Fondazione g. Pascale;s.c. Ematologia Oncologica, Napoli, Campania
  - Nuovo Policlinico, Ii Facolta; Divisione Di Ematologia, Napoli, Campania
  - Ospedale "A.Tortora" - Ematologia; Dipartimento Di Ematologia, Pagani (Sa), Campania
  - A.O. Universitaria Policlinico S.Orsola-Malpighi Di Bologna, Bologna, Emilia-Romagna
  - AUSL - IRCCS Santa Maria Nuova; U.O. Day Hospital di Oncologia, Reggio Emilia, Emilia-Romagna
  - A.O. Universitaria S. Maria Della Misericordia Di Udine; Oncologia; Clinica Ematologica, Udine, Friuli Venezia Giulia
  - Universita' Degli Studi La Sapienza-Ist.Di Ematologia; Dip Biot Cel e Ematol, Rome, Lazio
  - A.O. Universitaria S. Martino Di Genova; Ematologia 1, Genoa, Liguria
  - A.O. Spedali Civili Di Brescia-P.O. Spedali Civili;U.O. Ematologia, Brescia, Lombardy
  - Hospital San Raffaele, Milan, Lombardy
  - Ist. Nazionale Per Lo Studio E Cura Dei Tumori; Div. Ematologia Trapianto Midollo Osseo Allogenico, Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO); Emato-Oncologia, Milan, Lombardy
  - Irccs Policlinico San Matteo; Divisione Di Ematologia, Pavia, Lombardy
  - Ospedale Civile SS. Antonio E Biagio DI Alessandria; Ematologia, Alessandria, Piedmont
  - Ospedali Riuniti del Canavese, Ivrea, Piedmont
  - Univ. Piemonte Est Amedeo Avogadro; Div.Ematologia- Dip.Clinica Med.Sperim.& Ircad, Novara, Piedmont
  - Az. Osp. S. Luigi Gonzaga; S.C.D.U. Medicina Interna Ii, Orbassano, Piedmont
  - A.O. Universitaria S. Giovanni Battista-Molinette Di Torino; Ematologia 1, Turin, Piedmont
  - A.O.U. Citta' Della Salute E Della Scienza-P.O. Molinette;S.C. Ematologia, Turin, Piedmont
  - Azienda Ospedaliero Univ, Catania, Sicily
  - Az. Osp. Papardo; Struttura Complessa Di Ematologia, Messina, Sicily
  - Azienda Ospedaliera Univ, Florence, Tuscany
  - Ospedale Santa Chiara; Unita Operativa Di Ematologia, Pisa, Tuscany
  - Az. Osp. S. Maria; Dept. Di Oncologia Medica, Terni, Umbria
  - Ospedale Ca Foncello; Ematologia, Treviso, Veneto
  - Uni Di Verona Policlinico G.B. Rossi; Divisione E Cattedra Di Ematologia, Verona, Veneto
  - Ospedale Di Vicenza; Nefrologia, Ematologia, Vicenza, Veneto
- Japan (21):
  - Nagoya Daini Red Cross Hospital; Hematology & Oncology, Aichi
  - Chiba University Hospital; Hematology, Chiba
  - Kyushu University Hospital; Hematology, Oncology & Cardiovascular medicine, Fukuoka
  - Kurume University Hospital; Hematology and Oncology, Fukuoka
  - Gifu University Hospital; First Department of Internal Medicine, Gifu
  - Hokkaido University Hospital; Hematology, Hokkaido
  - Kobe City Medical Center General Hospital; Hematology, Hyōgo
  - Yokohama City University Hospital; Hematology, Rheumatology, Infectious Disease, Kanagawa
  - Kyoto University Hospital; Department of Hematology/Oncology, Kyoto
  - Niigata Cancer Center Hospital; Internal Medicine, Niigata
  - Iwate Medical University Hospital;Hematology and Oncology, Numakunai
  - Kurashiki Central Hospital; Hematology, Okayama
  - Osaka City University Hospital; Hematology, Osaka
  - Osaka University Hospital; Hematology and Oncology, Osaka
  - Kindai University Hospital; Hematology and Rheumatology, Osaka
  - Shimane University Hospital;Hematology, Shimane
  - Jichi Medical University Hospital; Hematology, Tochigi
  - National Cancer Center Hospital; Hematology, Tokyo
  - Toranomon Hospital; Hematology, Tokyo
  - Nippon Medical School Hospital; Hematology, Tokyo
  - The Cancer Institute Hospital of JFCR; Hematology Oncology, Tokyo
- Mexico (4):
  - Centro Estatal De Cancerologia De Chihuahua; Servicio De Hematologia Banco De Sangre, Chihuahua City
  - Hospital Universitario Dr. Jose E. Gonzalez; Haematology, Monterrey
  - Oaxaca Site Management Organization, Oaxaca City
  - Centro de Estudios Clinicos de Queretaro, SC, Querétaro
- Centro Hemato Oncologico Panama, Panama City, Panama
- Peru (3):
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
  - Instituto;Oncologico Miraflores, Lima
  - Clinica de Especialidades Medicas, Lima
- Poland (6):
  - Szpital Specjalistyczny Podkarpacki Ośrodek Onkologiczny, Brzozów
  - Uniwersyteckie Centrum Kliniczne; Klinika Hematologii i Transplantologii, Gdansk
  - Medical University of Lodz; Hematology, Lodz
  - Katedra i Klinika Hematoonkologii i Transplantacji Szpiku; Uniwersytetu Medycznego w Lublinie, Lublin
  - Centrum Onkologii Instytut im. M. Sklodowskiej-Curie, Klinika Nowotworow Ukladu Chlonnego, Warsaw
  - Medical Uni of Wroclaw; Hematology, Wroclaw
- Russia (6):
  - Clinical Oncology Dispensary of Ministry of Health of Tatarstan, Kazan'
  - Blokhin Cancer Research Center; Clinical Oncology, Moscow
  - Regional Clinical Hospital N.A. Semashko; Hematology, Nizhny Novgorod
  - Penza Regional Oncology Dispensary, Penza
  - Republican Clinical Hospital n.a. Baranov; Haematology, Petrozavodsk
  - Research Inst. of Hematology & Blood Transfusion ; Hematology, Saint Petersburg
- Serbia (2):
  - Institute of Hematology, Belgrade
  - Clinical Center Vojvodine; Clinic for Hematology, Novi Sad
- National Oncology Inst. ; Dept. of Haematology, Bratislava, Slovakia
- South Africa (5):
  - Constantiaberg Medical Clinic; Dept. of Haematology & Bone Marrow Translant, Cape Town
  - Mary Potter Oncology Centre, Groenkloof
  - Medical Oncology Centre of Rosebank; Oncology, Johannesburg
  - Wits Donald Gordon Clinical Trial Centre; Medical Oncology, Parktown, Johannesburg
  - Drs Thomson, Brittain an Partners Inc, Pretoria
- South Korea (7):
  - National Cancer Center, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Hospital, Seoul
  - Asan Medical Center - Oncology, Seoul
  - Yonsei University Severance Hospital; Medical Oncology, Seoul
  - St. Mary'S Hospital, the Catholic University School of Medicine; Internal Medicine, Seoul
  - Samsung Medical Center, Seoul
- Spain (10):
  - Hospital de Navarra, Servicio de Hematología, Pamplona, Navarre
  - Hospital Universitari Sant Joan de Reus; Servicio de Oncologia, Reus, Tarragona
  - Hospital del Mar; Servicio de Hematologia, Barcelona
  - Hospital Universitari Vall d'Hebron; Servicio de Hematologia, Barcelona
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Hospital Duran i Reynals; Servicio de Hematologia, Barcelona
  - Hospital Ramon y Cajal; Servicio de Hematologia, Madrid
  - Complejo Hospitalario de Pontevedra; Servicio de Oncologia, Pontevedra
  - Hospital Universitario Virgen Macarena; Servicio de Oncologia, Seville
  - Complejo Hospitalario de Toledo- H. Virgen de la Salud; Servicio de Oncologia, Toledo
- Switzerland (4):
  - Kantonsspital Aarau; Zentrum Für Onkologie, Hämatologie & Transfusionsmedizin, Aarau
  - Ospedale San Giovanni; Oncologia, Bellinzona
  - Kantonsspital Graubünden;Onkologie und Hämatologie, Chur
  - UniversitätsSpital Zürich; Zentrum für Hämatologie und Onkologie, Klinik für Onkologie, Zurich
- Taiwan (4):
  - Veterans General Hospital; Division of Oncology, Taipei
  - National Taiwan Universtiy Hospital; Division of Hematology, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center; Hemato-Oncology, Taipei
  - Chang Gung Medical Foundation - Linkou; Division of Hematology- Oncology, Taoyuan District
- Thailand (6):
  - King Chulalongkorn Memorial Hospital; Division of Hematology, Department of Medicine, Bangkok
  - National Cancer Inst., Bangkok
  - Rajavithi Hospital; Medicine, Bangkok
  - Ramathibodi Hospital; Division of Hematology, Department of Medicine, Bangkok
  - Siriraj Hospital; Division of Hematology, Department of Medicine, Bangkok
  - Srinagarind Hospital, Khon Kaen Uni ; Dept of Medicine, Khon Kaen
- United Kingdom (5):
  - Aberdeen Royal Infirmary; Haematology - Ward 16, Aberdeen
  - Birmingham Heartlands Hospital; Department of Haematology, Birmingham
  - Addenbrookes Hospital; Haematology, Cambridge
  - The HOPE Clinical Trials Unit, Leicester
  - New Cross Hospital; Dept. Of Haematology, Wolverhampton

REFERENCES:
- [Derived] Torkaman M, Jemaa S, Fredrickson J, Fernandez Coimbra A, De Crespigny A, Carano RAD. Comparative analysis of intestinal tumor segmentation in PET CT scans using organ based and whole body deep learning. BMC Med Imaging. 2025 Feb 17;25(1):52. doi: 10.1186/s12880-025-01587-3. PMID 39962481
- [Derived] Jemaa S, Ounadjela S, Wang X, El-Galaly TC, Kostakoglu L, Knapp A, Ku G, Musick L, Sahin D, Wei MC, Yin S, Bengtsson T, De Crespigny A, Carano RAD. Automated Lugano Metabolic Response Assessment in 18F-Fluorodeoxyglucose-Avid Non-Hodgkin Lymphoma With Deep Learning on 18F-Fluorodeoxyglucose-Positron Emission Tomography. J Clin Oncol. 2024 Sep 1;42(25):2966-2977. doi: 10.1200/JCO.23.01978. Epub 2024 Jun 6. PMID 38843483
- [Derived] Yan JT, Bel C, Trask PC, Lo E. Are changes in patient-reported outcomes prognostic for diffuse large B-Cell lymphoma survival? Results from the GOYA trial. J Patient Rep Outcomes. 2024 Mar 18;8(1):31. doi: 10.1186/s41687-024-00708-w. PMID 38498084
- [Derived] Ho RS, Launonen A. Comparison of statistical methods for extrapolating survival in previously untreated diffuse large B-cell lymphoma: results based on the POLARIX study. J Med Econ. 2023 Jan-Dec;26(1):1178-1189. doi: 10.1080/13696998.2023.2259107. Epub 2023 Sep 13. PMID 37702406
- [Derived] Jemaa S, Paulson JN, Hutchings M, Kostakoglu L, Trotman J, Tracy S, de Crespigny A, Carano RAD, El-Galaly TC, Nielsen TG, Bengtsson T. Full automation of total metabolic tumor volume from FDG-PET/CT in DLBCL for baseline risk assessments. Cancer Imaging. 2022 Aug 12;22(1):39. doi: 10.1186/s40644-022-00476-0. PMID 35962459
- [Derived] Nowicka M, Hilton LK, Ashton-Key M, Hargreaves CE, Lee C, Foxall R, Carter MJ, Beers SA, Potter KN, Bolen CR, Klein C, Knapp A, Mir F, Rose-Zerilli M, Burton C, Klapper W, Scott DW, Sehn LH, Vitolo U, Martelli M, Trneny M, Rushton CK, Slack GW, Farinha P, Strefford JC, Oestergaard MZ, Morin RD, Cragg MS. Prognostic significance of FCGR2B expression for the response of DLBCL patients to rituximab or obinutuzumab treatment. Blood Adv. 2021 Aug 10;5(15):2945-2957. doi: 10.1182/bloodadvances.2021004770. PMID 34323958
- [Derived] Strefford JC, Nowicka M, Hargreaves CE, Burton C, Davies A, Ganderton R, Hiddemann W, Iriyama C, Klapper W, Latham KV, Martelli M, Mir F, Parker H, Potter KN, Rose-Zerilli MJJ, Sehn LH, Trneny M, Vitolo U, Bolen CR, Klein C, Knapp A, Oestergaard MZ, Cragg MS. Single-nucleotide Fcgamma receptor polymorphisms do not impact obinutuzumab/rituximab outcome in patients with lymphoma. Blood Adv. 2021 Aug 10;5(15):2935-2944. doi: 10.1182/bloodadvances.2020003985. PMID 34323957
- [Derived] Kostakoglu L, Martelli M, Sehn LH, Belada D, Carella AM, Chua N, Gonzalez-Barca E, Hong X, Pinto A, Shi Y, Tatsumi Y, Knapp A, Mattiello F, Nielsen T, Sahin D, Sellam G, Oestergaard MZ, Vitolo U, Trneny M. End-of-treatment PET/CT predicts PFS and OS in DLBCL after first-line treatment: results from GOYA. Blood Adv. 2021 Mar 9;5(5):1283-1290. doi: 10.1182/bloodadvances.2020002690. PMID 33651099
- [Derived] Bolen CR, Klanova M, Trneny M, Sehn LH, He J, Tong J, Paulson JN, Kim E, Vitolo U, Di Rocco A, Fingerle-Rowson G, Nielsen T, Lenz G, Oestergaard MZ. Prognostic impact of somatic mutations in diffuse large B-cell lymphoma and relationship to cell-of-origin: data from the phase III GOYA study. Haematologica. 2020 Sep 1;105(9):2298-2307. doi: 10.3324/haematol.2019.227892. PMID 33054054
- [Derived] Sehn LH, Martelli M, Trneny M, Liu W, Bolen CR, Knapp A, Sahin D, Sellam G, Vitolo U. A randomized, open-label, Phase III study of obinutuzumab or rituximab plus CHOP in patients with previously untreated diffuse large B-Cell lymphoma: final analysis of GOYA. J Hematol Oncol. 2020 Jun 6;13(1):71. doi: 10.1186/s13045-020-00900-7. PMID 32505213
- [Derived] Klanova M, Oestergaard MZ, Trneny M, Hiddemann W, Marcus R, Sehn LH, Vitolo U, Bazeos A, Goede V, Zeuner H, Knapp A, Sahin D, Spielewoy N, Bolen CR, Cardona A, Klein C, Venstrom JM, Nielsen T, Fingerle-Rowson G. Prognostic Impact of Natural Killer Cell Count in Follicular Lymphoma and Diffuse Large B-cell Lymphoma Patients Treated with Immunochemotherapy. Clin Cancer Res. 2019 Aug 1;25(15):4634-4643. doi: 10.1158/1078-0432.CCR-18-3270. Epub 2019 May 3. PMID 31053601
- [Derived] McCord R, Bolen CR, Koeppen H, Kadel EE 3rd, Oestergaard MZ, Nielsen T, Sehn LH, Venstrom JM. PD-L1 and tumor-associated macrophages in de novo DLBCL. Blood Adv. 2019 Feb 26;3(4):531-540. doi: 10.1182/bloodadvances.2018020602. PMID 30770362
- [Derived] Klanova M, Sehn LH, Bence-Bruckler I, Cavallo F, Jin J, Martelli M, Stewart D, Vitolo U, Zaja F, Zhang Q, Mattiello F, Sellam G, Punnoose EA, Szafer-Glusman E, Bolen CR, Oestergaard MZ, Fingerle-Rowson GR, Nielsen T, Trneny M. Integration of cell of origin into the clinical CNS International Prognostic Index improves CNS relapse prediction in DLBCL. Blood. 2019 Feb 28;133(9):919-926. doi: 10.1182/blood-2018-07-862862. Epub 2019 Jan 7. PMID 30617197
- [Derived] Kusumoto S, Arcaini L, Hong X, Jin J, Kim WS, Kwong YL, Peters MG, Tanaka Y, Zelenetz AD, Kuriki H, Fingerle-Rowson G, Nielsen T, Ueda E, Piper-Lepoutre H, Sellam G, Tobinai K. Risk of HBV reactivation in patients with B-cell lymphomas receiving obinutuzumab or rituximab immunochemotherapy. Blood. 2019 Jan 10;133(2):137-146. doi: 10.1182/blood-2018-04-848044. Epub 2018 Oct 19. PMID 30341058

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1418 patients were randomized and included in the primary analyses (29 April 2016). A total of 1414 patients were included in the final analysis (31 January 2018), 710 in the R-CHOP arm and 704 in the G-CHOP arm; data from 4 patients were excluded because of serious GCP non-compliance at a single study site in China.
Period: Overall Study
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Started | 712 | 706
Completed | 86 | 91
Not Completed | 626 | 615
Not completed — Withdrawal by Subject | 35 | 38
Not completed — Protocol Violation | 2 | 0
Not completed — Physician Decision | 15 | 23
Not completed — Non-compliance | 8 | 6
Not completed — Lost to Follow-up | 10 | 8
Not completed — Death | 32 | 44
Not completed — Adverse Event | 4 | 6
Not completed — Study terminated by Sponsor | 307 | 315
Not completed — Progressive disease | 190 | 166
Not completed — Reason not specified | 23 | 9

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all randomized participants. However, 4 patients were classified as misconduct patients and were not included in the ITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy | Total
Number analyzed (Participants) | 710 | 704 | 1414
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (13.6) | 59.4 (13.3) | 59.2 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 328 | 336 | 664
  Male | 382 | 368 | 750

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Progression-Free Survival (PFS), Investigator-Assessed
Description: Kaplan Meier estimate of the median PFS was defined as the time at which half of the participants have progressed (progressive disease [PD]). Progression-free survival was defined as the time from randomization until the first documented day of disease progression or relapse, using a modified version of the Revised Response Criteria for Malignant Lymphoma, or death from any cause, whichever occurred first, on the basis of investigator assessments. Progression was defined as at least 50% increase in nodal lesions or >/=50% increase in any node > 1 centimeter (cm) or >/= 50% increase in other target measurable lesions (e.g., splenic or hepatic nodules) and/or appearance of any new bone marrow involvement and/or appearance of any new lesion > 1.5 cm or >/= 50% increase in any previously involved node with a diameter </= 1 cm such that it is now >1.5 cm. Tumor measurements were obtained by computed tomography (CT) or magnetic resonance imaging (MRI).
Time Frame: Baseline up to approximately 6.5 years (up to 31 January 2018)
Population: The intent-to-treat (ITT) population included all randomized participants, however because of serious Good Clinical Practice non-compliance at a single study site in China, all 4 participants enrolled at the site (2 in each treatment arm) were excluded from the final analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 710 | 704
months | 74.5 [NA to NA] — The 95% CI could not be estimated as too few participants had an event. | 68.3 [68.3 to NA] — Upper bound of 95% CI could not be estimated as too few participants had an event.
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Test type: Superiority or Other; p = 0.4753, Log Rank; Stratified by International Prognostic Index (IPI) score (low/low-intermediate (excluding participants having an IPI score 0 without bulky disease); Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.78 to 1.12]

2. Secondary Outcome: Median Time to Progression-Free Survival (PFS), Independent Review Committee (IRC)-Assessed
Description: Kaplan Meier estimate of median PFS was defined as time at which half of participants have progressed (progressive disease [PD]). Progression-free survival was defined as time from randomization until first documented day of disease progression or relapse, using a modified version of Revised Response Criteria for Malignant Lymphoma, or death from any cause, whichever occurred first, on basis of IRC assessments. Progression was defined as at least 50% increase in nodal lesions or >/=50% increase in any node > 1 cm or >/= 50% increase in other target measurable lesions (e.g., splenic or hepatic nodules) and/or appearance of any new bone marrow involvement and/or appearance of any new lesion > 1.5 cm or >/= 50% increase in any previously involved node with diameter </= 1 cm such that it is now >1.5 cm. Tumor measurements were obtained by CT or MRI. This outcome measure used data from primary analysis which included all 1418 participants.
Time Frame: Baseline up to approximately 4 years and 9 months (up to 29 April 2016)
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 712 | 706
months | NA [NA to NA] — Median and corresponding 95% CI could not be estimated as too few participants had an event. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated as too few participants had an event.
Statistical Analysis 1: Comparison: Rituximab+Chemotherapy vs Obinutuzumab+Chemotherapy; Test type: Superiority or Other; p = 0.2736, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.72 to 1.10]

3. Secondary Outcome: Median Time to Overall Survival (OS)
Description: Kaplan Meier estimate of median OS was defined as the time at which half of the participants had died, regardless of the cause of death. Overall survival in the overall study population was defined as the time from the date of randomization to the date of death from any cause.
Time Frame: Baseline up to approximately 6.5 years (up to 31 January 2018)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 710 | 704
months | NA [NA to NA] — Median and corresponding 95% CI could not be estimated as too few participants had an event. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated as too few participants had an event.

4. Secondary Outcome: Overall Response Rate (ORR), Investigator-Assessed
Description: Overall response was determined on the basis of investigator assessments according to the International Working Group (IWG) Revised Response Criteria for Malignant Lymphoma, 2007. Tumor assessments were performed with CT/MRI with or without PET. Overall response was defined as the disappearance of all evidence of disease, regression of measurable disease, and no new sites.
Time Frame: Baseline up to approximately 6.5 years (up to 31 January 2018)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 710 | 704
percentage of participants
  Without PET | 80.1 | 81.4
  With PET: number analyzed (Participants) | 665 | 669
  With PET | 77.6 | 77.1

5. Secondary Outcome: Overall Response Rate (ORR), IRC-Assessed
Description: Overall response was determined on the basis of IRC assessments according to the International Working Group (IWG) Revised Response Criteria for Malignant Lymphoma, 2007. Tumor assessments were performed with CT/MRI with or without PET. Overall response was defined as the disappearance of all evidence of disease, regression of measurable disease, and no new sites. This outcome measure used data from primary analysis which included all 1418 participants.
Time Frame: Baseline up to approximately 4 years and 9 months (up to 29 April 2016)
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 712 | 706
percentage of participants
  Without PET | 80.2 | 82.3
  With PET: number analyzed (Participants) | 665 | 669
  With PET | 81.1 | 82.1

6. Secondary Outcome: Complete Response (CR) at the End of Treatment, Investigator-Assessed
Description: Percentage of participants with complete response was determined on the basis of investigator assessments according to the International Working Group (IWG) Revised Response Criteria for Malignant Lymphoma, 2007. Tumor assessments were performed with CT/MRI with or without PET. Complete response was defined as the disappearance of all evidence of disease.
Time Frame: Baseline up to approximately 6.5 years (up to 31 January 2018)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 710 | 704
percentage of participants
  Without PET | 33.9 | 35.4
  With PET: number analyzed (Participants) | 665 | 669
  With PET | 59.1 | 56.5

7. Secondary Outcome: Complete Response (CR) at the End of Treatment, IRC-Assessed
Description: Percentage of participants with complete response was determined on the basis of IRC assessments according to the International Working Group (IWG) Revised Response Criteria for Malignant Lymphoma, 2007. Tumor assessments were performed with CT/MRI with or without PET. Complete response was defined as the disappearance of all evidence of disease. This outcome measure used data from primary analysis which included all 1418 participants.
Time Frame: Baseline up to approximately 4 years and 9 months (up to 29 April 2016)
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 712 | 706
percentage of participants
  Without PET | 34.4 | 39.1
  With PET: number analyzed (Participants) | 665 | 669
  With PET | 65.3 | 66.7

8. Secondary Outcome: Median Time to Event-Free Survival (EFS), Investigator-Assessed
Description: Kaplan Meier estimate of median EFS is the time at which half of the participants have progressed. Event-free survival was defined as the time from the date of randomization until the date of disease progression, relapse, initiation of a new non-protocol-specified anti-lymphoma treatment, or death from any cause on the basis of investigator assessments with the use of Revised Response Criteria for Malignant Lymphoma. Disease progression/relapse was defined as at least 50% increase in nodal lesions or >/=50% increase in any node > 1 centimeter (cm) or >/= 50% increase in other target measurable lesions (e.g., splenic or hepatic nodules) and/or appearance of any new bone marrow involvement and/or appearance of any new lesion > 1.5 cm or >/= 50% increase in any previously involved node with a diameter </= 1 cm such that it is now >1.5 cm. Tumor measurements were obtained by CT/MRI.
Time Frame: Baseline up to death or disease progression, or initiation of new anti-lymphoma treatment (NALT), whichever occurred first, approximately 6.5 years (up to 31 January 2018)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 710 | 704
months | 74.5 [NA to NA] — The 95% CI could not be estimated as too few participants had an event. | 68.3 [68.3 to NA] — The upper bound of 95% CI could not be estimated as too few participants had an event.

9. Secondary Outcome: Median Time to Disease-Free Survival (DFS), Investigator-Assessed
Description: Kaplan Meier estimate of median DFS was defined as time at which half of participants have disease progression/relapse or death from any cause. Disease-free survival was defined as time from date of the first occurrence of a documented CR to date of disease progression/relapse or death from any cause on basis of investigator assessments with use of Revised Response Criteria for Malignant Lymphoma. Tumor assessments were performed with CT/MRI. CR was defined as disappearance of all target lesions. Progression/relapse was defined as at least 50% increase in nodal lesions or >/=50% increase in any node > 1 centimeter (cm) or >/= 50% increase in other target measurable lesions (e.g., splenic or hepatic nodules) and/or appearance of any new bone marrow involvement and/or appearance of any new lesion > 1.5 cm or >/= 50% increase in any previously involved node with a diameter </= 1 cm such that it is now >1.5 cm.
Time Frame: Baseline up to death or disease progression, whichever occurred first, approximately 6.5 years (up to 31 January 2018)
Population: The intent-to-treat (ITT) population included all randomized participants, of which evaluable participants were included in this analysis, however because of serious Good Clinical Practice non-compliance at a single study site in China, all 4 participants enrolled at the site (2 in each treatment arm) were excluded from the final analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 394 | 417
months | NA [NA to NA] — Median and corresponding 95% CI could not be estimated as too few participants had an event. | 65.4 [NA to NA] — The 95% CI could not be estimated as too few participants had an event.

10. Secondary Outcome: Duration of Response (DOR), Investigator-Assessed
Description: DOR: time from first occurrence of documented CR or PR to disease progression/relapse, or death from any cause for participants with a response of CR or PR. Tumor assessments were performed with CT/MRI. CR: disappearance of all target lesions. PR: >/=50% decrease target lesions in up to six dominant lesions identified at baseline, no new lesions and no increase in the size of the liver, spleen, or other nodes. Splenic and hepatic nodule regression >/= 50%. Progression/relapse: at least 50% increase in nodal lesions or >/=50% increase in any node > 1 cm or >/= 50% increase in other target lesions (e.g., splenic or hepatic nodules) and/or any new bone marrow involvement and/or any new lesion > 1.5 cm or >/= 50% increase in any previously involved node with a diameter </= 1 cm such that it is now >1.5 cm. A participant in the Rituximab+CHOP arm with the longest follow-up, 53 months, had an event. The criterion for median was the minimum time when survival went below 50%.
Time Frame: Baseline up to death or disease progression, whichever occurred first, approximately 6.5 years (up to 31 January 2018)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 641 | 657
months | 71.9 [NA to NA] — There were not enough events to calculate the confidence intervals. | NA [65.4 to NA] — There were not enough events to calculate the median and the upper limit of the confidence interval.

11. Secondary Outcome: Time to Next Anti-Lymphoma Treatment (TTNALT)
Description: Time to next anti-lymphoma treatment was defined as the time from the date of randomization to the start date of the next anti-lymphoma treatment or death from any cause.
Time Frame: Baseline up to start of next anti-lymphoma treatment or death due to any cause, whichever occurred first, approximately 6.5 years (31 January 2018)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 710 | 704
months | NA [74.5 to NA] — Median and upper limit of the 95% confidence interval were not calculable, due to too few participants had an event. | NA [NA to NA] — Median and 95% confidence interval were not calculable, due to too few participants had an event.

12. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up to approximately 6.5 years (up to 31 January 2018)
Population: The safety analysis population included all participants who received at least one dose of study drug. Because of serious Good Clinical Practice non-compliance at a single study site in China, all 4 participants enrolled at the site (2 in each treatment arm) were excluded from the final analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 701 | 702
percentage of participants | 95.3 | 98.1

13. Secondary Outcome: Percentage of Participants With Human Anti-Human Antibodies (HAHAs) to Obinutuzumab
Description: The presence of HAHAs to obinutuzumab was assessed in the first 100 randomized participants.
Time Frame: Pre-dose (Hour 0) on Cycle (C) 4 Day (D) 1, at end of treatment/early termination (up to Month 6), every 6 months thereafter for 30 months (cycle length = 21 days)
Population: The safety analysis population included all participants who received at least one dose of study drug. Because of serious Good Clinical Practice non- compliance at a single study site in China, all 4 participants enrolled at the site (2 in each treatment arm) were excluded from the final analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 100
percentage of participants
  Screening | 2.0
  Cycle 4 Day 1: number analyzed (Participants) | 86
  Cycle 4 Day 1 | 0
  Study Completion / Early Discontinuation: number analyzed (Participants) | 65
  Study Completion / Early Discontinuation | 0
  Follow-Up Month 6: number analyzed (Participants) | 40
  Follow-Up Month 6 | 0
  Follow-Up Month 12: number analyzed (Participants) | 40
  Follow-Up Month 12 | 0
  Follow-Up Month 18: number analyzed (Participants) | 27
  Follow-Up Month 18 | 0
  Follow-Up Month 24: number analyzed (Participants) | 25
  Follow-Up Month 24 | 0
  Follow-Up Month 30: number analyzed (Participants) | 19
  Follow-Up Month 30 | 0
  Follow-Up Completion/ Early Discontinuation: number analyzed (Participants) | 46
  Follow-Up Completion/ Early Discontinuation | 0
  Unscheduled: number analyzed (Participants) | 3
  Unscheduled | 0

14. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym) Subscale Score
Description: The FACT-Lym subscale was developed to assess health-related quality of life in participants with non-Hodgkin lymphoma. The score range is 0-60, with higher scores indicating better outcomes. A positive change from baseline indicates an improvement.
Time Frame: Baseline (pre-dose [Hour 0] on C1D1), C3D1, end of treatment (up to Month 6), every 12 months thereafter up to approximately 6.5 years, (cycle length = 21 days)
Population: The intent-to-treat (ITT) population included all randomized participants. Because of serious Good Clinical Practice non-compliance at a single study site in China, all 4 participants enrolled at the site (2 in each treatment arm) were excluded from the final analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 710 | 706
score on a scale
  Baseline: number analyzed (Participants) | 609 | 639
  Baseline | 45.34 (10.16) | 45.18 (9.86)
  Score Change, Cycle 3 Day 1: number analyzed (Participants) | 553 | 563
  Score Change, Cycle 3 Day 1 | 3.83 (8.65) | 3.70 (9.13)
  Score Change, Study Compl./Discont.: number analyzed (Participants) | 526 | 527
  Score Change, Study Compl./Discont. | 5.03 (10.21) | 4.35 (11.03)
  Score Change, Follow-Up Month 12: number analyzed (Participants) | 371 | 411
  Score Change, Follow-Up Month 12 | 6.37 (10.12) | 6.18 (10.51)
  Score Change, Follow-Up Month 24: number analyzed (Participants) | 335 | 372
  Score Change, Follow-Up Month 24 | 7.07 (10.35) | 6.66 (10.50)
  Score Change, Follow-Up Month 30: number analyzed (Participants) | 0 | 1
  Score Change, Follow-Up Month 30 |  | 25.00 (NA) — NA = NE = Not estimable based on 1 participant evaluated
  Score Change, Follow-Up Month 36: number analyzed (Participants) | 317 | 353
  Score Change, Follow-Up Month 36 | 7.57 (10.16) | 7.31 (10.67)
  Score Change, Follow-Up Month 48: number analyzed (Participants) | 167 | 192
  Score Change, Follow-Up Month 48 | 8.22 (9.65) | 7.37 (10.45)
  Score Change, Follow-Up Term./Compl.: number analyzed (Participants) | 121 | 135
  Score Change, Follow-Up Term./Compl. | 5.51 (10.04) | 5.55 (10.62)

15. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Core 30 (EORTC QLQ-C30) Domain Scores
Description: The EORTC QLQ-C30 is a health-related quality of life questionnaire. A higher score indicates better quality of life, with changes of 5 to 10 points considered to be a minimally important difference to participants.
Time Frame: Baseline (pre-dose [Hour 0] on C1D1), C3D1, end of treatment (up to Month 6), every 12 months thereafter up to data cut-off, up to approximately 6.5 years, (cycle length = 21 days)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 710 | 704
score on a scale
  Baseline: number analyzed (Participants) | 610 | 641
  Baseline | 59.81 (24.39) | 58.55 (25.23)
  Change Baseline, Cycle 1 Day 1: number analyzed (Participants) | 0 | 0
  Change Baseline, Cycle 3 Day 1: number analyzed (Participants) | 556 | 565
  Change Baseline, Cycle 3 Day 1 | 6.37 (23.77) | 7.51 (25.99)
  Change Baseline, Study Completion: number analyzed (Participants) | 526 | 530
  Change Baseline, Study Completion | 9.84 (25.96) | 10.22 (30.17)
  Change Baseline, Follow-Up Month 12: number analyzed (Participants) | 371 | 413
  Change Baseline, Follow-Up Month 12 | 12.67 (26.31) | 13.84 (29.97)
  Change Baseline, Follow-Up Month 24: number analyzed (Participants) | 337 | 370
  Change Baseline, Follow-Up Month 24 | 14.74 (26.33) | 15.81 (29.24)
  Change Baseline, Follow-Up Month 30: number analyzed (Participants) | 0 | 1
  Change Baseline, Follow-Up Month 30 |  | 58.33 (NA) — NA = NE = Not estimable based on 1 participant evaluated
  Change Baseline, Follow-Up Month 36: number analyzed (Participants) | 321 | 352
  Change Baseline, Follow-Up Month 36 | 15.01 (26.85) | 17.99 (28.85)
  Change Baseline, Follow-Up Month 48: number analyzed (Participants) | 168 | 193
  Change Baseline, Follow-Up Month 48 | 16.62 (27.49) | 17.53 (30.31)
  Change Baseline, Follow-Up Completion: number analyzed (Participants) | 122 | 136
  Change Baseline, Follow-Up Completion | 8.74 (29.40) | 8.46 (28.71)

16. Secondary Outcome: Serum Concentrations of Obinutuzumab in Japanese Participants With Diffuse Large B-Cell Lymphoma (DLBCL)
Description: Serum samples for assessment of obinutuzumab serum concentrations were collected only from a subset of Japanese participants following administration of 1000 mg obinutuzumab.
Time Frame: C1: D1 post-infusion and 20-28 and 66-80 hours after end of infusion, D8 and D15 pre-and post-infusion; C2: D1 pre- and post-infusion; C4: D1 pre- and post-infusion; C6: D1 pre- and post-infusion; C8: D1 pre- and post-infusion (cycle length = 21 days)
Population: The Pharmacokinetic assessment was done on a subset of 39 Japanese participants in the Obinutuzumab+Chemotherapy arm only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Obinutuzumab+Chemotherapy
Number analyzed (Participants) | 39
micrograms per milliliter (μg/mL)
  Cycle 1, Day 8 pre-infusion | 174 (38.7)
  Cycle 1, Day 15 pre-infusion | 320 (39.2)
  Cycle 2, Day 1 pre-infusion | 431 (39.8)
  Cycle 4, Day 1 pre-infusion | 352 (42.1)
  Cycle 6, Day 1 pre-infusion | 378 (45.9)
  Cycle 8, Day 1 pre-infusion | 478 (43.9)
  Cycle 1, Day 1 post-infusion | 435 (32.3)
  Cycle 1, Day 1 20-28 hours after end of infusion | 259 (56.3)
  Cycle 1, Day 1 66-80 hours after end of infusion | 219 (51.2)
  Cycle 1, Day 8 post-infusion | 578 (37.8)
  Cycle 1, Day 15 post-infusion | 718 (32.9)
  Cycle 2, Day 1 post-infusion | 938 (31.3)
  Cycle 4, Day 1 post-infusion | 817 (28.6)
  Cycle 6, Day 1 post-infusion | 813 (32.6)
  Cycle 8, Day 1 post-infusion | 881 (35.9)

ADVERSE EVENTS:
Time Frame: 6 years and 7 months
Description: The safety analysis population included all participants who received at least one dose of study drug (i.e., obinutuzumab, rituximab, or CHOP). Because of serious Good Clinical Practice non-compliance at a single study site in China, all 4 patients enrolled at the site (2 in each treatment arm) were excluded from the final analysis.
Arm/Group | Rituximab+Chemotherapy | Obinutuzumab+Chemotherapy
Serious Adverse Events (participants affected / at risk) | 269/701 | 312/702
Other Adverse Events (participants affected / at risk) | 613/701 | 646/702
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab+Chemotherapy (N=701) | Obinutuzumab+Chemotherapy (N=702)
Anaemia (Blood and lymphatic system disorders) | 6 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 71 | 85
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 0 | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 6 | 14
Neutropenia (Blood and lymphatic system disorders) | 38 | 54
Splenic haematoma (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 12
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 5 | 2
Angina pectoris (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 9
Atrial flutter (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 3 | 7
Cardiac failure congestive (Cardiac disorders) | 1 | 3
Cardiac perforation (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary artery thrombosis (Cardiac disorders) | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Mitral valve disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 3
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular flutter (Cardiac disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Addison's disease (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 2 | 0
Lacrimation increased (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 4
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Anal fistula (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 5
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 1
Gastric perforation (Gastrointestinal disorders) | 3 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Ileal perforation (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 2 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 5 | 2
Intestinal perforation (Gastrointestinal disorders) | 3 | 3
Large intestine polyp (Gastrointestinal disorders) | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Small intestinal perforation (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 4 | 2
Axillary pain (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 0
Chills (General disorders) | 1 | 2
Death (General disorders) | 2 | 3
Extravasation (General disorders) | 1 | 0
Fatigue (General disorders) | 5 | 4
General physical health deterioration (General disorders) | 1 | 2
Hernia (General disorders) | 0 | 1
Hyperpyrexia (General disorders) | 0 | 1
Incarcerated hernia (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 2
Mucosal inflammation (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 11 | 17
Sudden death (General disorders) | 1 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 2
Appendiceal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 3 | 1
Atypical pneumonia (Infections and infestations) | 2 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 4 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 1
Candida sepsis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 2
Cholecystitis infective (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 | 3
Cytomegalovirus colitis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 2 | 1
Device related sepsis (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 1
Enterobacter infection (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 2
H1N1 influenza (Infections and infestations) | 0 | 1
Hepatitis B Reactivation (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 2
Herpes zoster (Infections and infestations) | 3 | 4
Herpes zoster disseminated (Infections and infestations) | 0 | 1
Infected lymphocele (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 2
Infectious pleural effusion (Infections and infestations) | 0 | 2
Infective glossitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 1
Laryngitis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 3
Lung infection (Infections and infestations) | 3 | 6
Measles (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Meningitis cryptococcal (Infections and infestations) | 1 | 0
Meningitis viral (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0
Neutropenic infection (Infections and infestations) | 1 | 1
Neutropenic sepsis (Infections and infestations) | 3 | 3
Oral infection (Infections and infestations) | 2 | 0
Orchitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 1
Peritonitis (Infections and infestations) | 2 | 2
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 33 | 43
Pneumonia bacterial (Infections and infestations) | 0 | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 1
Prostatic abscess (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 2
Scrotal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 10 | 16
Sepsis syndrome (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 3 | 12
Sinusitis fungal (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0
Tuberculosis of central nervous system (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 3 | 3
Urosepsis (Infections and infestations) | 1 | 1
Varicella (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 0 | 1
Viral pharyngitis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 8
Kidney rupture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 3
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
HIV antibody positive (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 4 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 2 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 3
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Embolic stroke (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 3
Hemiparesis (Nervous system disorders) | 0 | 1
Iiird nerve paralysis (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 2
Stroke in evolution (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Emotional distress (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 2
Cystitis glandularis (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 2
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 2
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 3
Orthostatic hypotension (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 2 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Venous occlusion (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
Bone Marrow Failure (Blood and lymphatic system disorders) | 1 | 0
Anorectal cellulitis (Infections and infestations) | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Angioimmuoblastic T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carincoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Axillary vein thrombosis (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Gastrointestinal Infection (Infections and infestations) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab+Chemotherapy (N=701) | Obinutuzumab+Chemotherapy (N=702)
Anaemia (Blood and lymphatic system disorders) | 101 | 96
Febrile neutropenia (Blood and lymphatic system disorders) | 44 | 52
Leukopenia (Blood and lymphatic system disorders) | 90 | 117
Neutropenia (Blood and lymphatic system disorders) | 269 | 315
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 58
Abdominal pain (Gastrointestinal disorders) | 47 | 47
Abdominal pain upper (Gastrointestinal disorders) | 41 | 38
Constipation (Gastrointestinal disorders) | 177 | 167
Diarrhoea (Gastrointestinal disorders) | 91 | 113
Dyspepsia (Gastrointestinal disorders) | 43 | 44
Nausea (Gastrointestinal disorders) | 199 | 210
Stomatitis (Gastrointestinal disorders) | 65 | 47
Vomiting (Gastrointestinal disorders) | 75 | 105
Asthenia (General disorders) | 74 | 76
Chills (General disorders) | 37 | 132
Fatigue (General disorders) | 124 | 136
Mucosal inflammation (General disorders) | 36 | 45
Oedema peripheral (General disorders) | 40 | 35
Pyrexia (General disorders) | 75 | 137
Upper respiratory tract infection (Infections and infestations) | 49 | 43
Infusion related reaction (Injury, poisoning and procedural complications) | 162 | 251
Decreased appetite (Metabolism and nutrition disorders) | 74 | 98
Hypokalaemia (Metabolism and nutrition disorders) | 55 | 67
Back pain (Musculoskeletal and connective tissue disorders) | 41 | 58
Dizziness (Nervous system disorders) | 29 | 48
Dysgeusia (Nervous system disorders) | 38 | 44
Headache (Nervous system disorders) | 58 | 75
Neuropathy peripheral (Nervous system disorders) | 88 | 87
Paraesthesia (Nervous system disorders) | 50 | 55
Peripheral sensory neuropathy (Nervous system disorders) | 57 | 54
Insomnia (Psychiatric disorders) | 61 | 79
Cough (Respiratory, thoracic and mediastinal disorders) | 66 | 88
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 | 52
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 38 | 43
Alopecia (Skin and subcutaneous tissue disorders) | 144 | 148
Rash (Skin and subcutaneous tissue disorders) | 45 | 17
Hypertension (Vascular disorders) | 27 | 40
Alanine Aminotransferase Increased (Investigations) | 29 | 39
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.